CLINICAL TRIAL: NCT02691962
Title: A Post-Market, Prospective, Multicenter, Single-Arm Trial of XenMatrix™ AB Surgical Graft in All Wound Classes Ventral or Incisional Midline Hernias
Brief Title: Xen Matrix™ AB Surgical Graft in Ventral or Incisional Midline Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVL-HE-012
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xen Matrix AB (Experimental): Subjects treated with Xen Matrix AB
  Interventions: Device: Xen Matrix AB

INTERVENTIONS:
Device: Xen Matrix AB — Xen Matrix™ AB Surgical Graft is an acellular, sterile, non-pyrogenic porcine dermal matrix packed dry for use in the reconstruction of soft tissue deficiencies. The device surfaces are coated with the antibacterial agents Rifampin and Minocycline in a bioresorbable L-Tyrosine succinate polymer carrier.

SUMMARY:
This study aims to prospectively explore the use of XenMatrix™ AB Surgical Graft for ventral or incisional midline hernia repair in patients across all wound classes ("All Comers") through 24 months post repair.

DETAILED DESCRIPTION:
This is a post-market, on-label study to understand the performance of the graft in the US.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing and able to give written informed consent.
* Subject must be diagnosed with a ventral or incisional midline hernia.
* Mesh must be placed in the retro-rectus or intraperitoneal plane.
* Subject must be willing to undergo open hernia repair and be able to undergo all other study procedures as outlined in this protocol.

Exclusion Criteria:

* The use of surgical graft as a bridge repair.
* The subject has more than 4 prior recurrences.
* Subject has a contraindication for the placement of surgical graft.
* Complete removal of existing mesh from a prior hernia repair (in the same affected area) is not possible.
* The study hernia repair requires more than a single piece mesh (including sufficient overlap beyond margins of the defect on all sides).
* Subject has intact permanent mesh adjacent to the current hernia to be repaired.
* Subject has peritonitis at the time of surgery.
* The subject is an active smoker within the last 2 weeks prior to surgery.
* Clinically significant Chronic Obstructive Pulmonary Disease or heart failure, defined as marked limitation in ability or inability to perform activities of daily living.
* Subject had chemotherapy within the last 12 months, is on or suspected to be placed on chemotherapy medications during any part of the study.
* Chronic steroid use (>6 months) or immunosuppression drugs.
* Subject's body mass index (BMI) >45 kg/m2.
* Subject has cirrhosis, and/or ascites.
* Subject has a defined collagen disorder.
* Known to be infected with human immunodeficiency virus (HIV).
* Subject has clinically significant (not based solely on creatinine levels) kidney disease that limits Activities of Daily Living, is on hemodialysis or peritoneal dialysis.
* Subject is American Society of Anesthesiology (ASA) Class 4 or 5.
* Subject has a life expectancy < 2 years at the time of enrollment.
* Subject is pregnant, breastfeeding or planning on becoming pregnant during the course of the study.
* Subjects with known sensitivity to porcine products.
* Subjects with allergy, history of allergy or hypersensitivity to tetracyclines (including minocycline) or rifamycins (including rifampin).
* Subject has any condition in the opinion of the Investigator that would preclude the use of the study device, or preclude the subject from completing the follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-05; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martindale, MD, Principal Investigator — Oregon Health and Science University
Locations (11):
- United States (11):
  - Keck Hospital of USC, Los Angeles, California
  - California Pacific Medical Center - Sutter Health, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Treated With Xen Matrix AB: This group includes participants with a diagnosis of ventral or incisional midline hernia who have undergone the hernia surgical repair with the use of the XenMatrix AB.
Period: Overall Study
Arm/Group | Subjects Treated With Xen Matrix AB
Started | 75
Completed | 59
Not Completed | 16

BASELINE CHARACTERISTICS:
Groups:
- Subjects Treated With XenMatrix AB: This group includes participants with a diagnosis of ventral or incisional midline hernia who have undergone the hernia surgical repair with the use of the XenMatrix AB.
Arm/Group | Subjects Treated With XenMatrix AB
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 60
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Occurrences Up to 45 Days Post Implantation
Description: Wound occurrences were defined as surgical site infection, seroma, wound dehiscence, skin necrosis and fistulas requiring intervention.
Time Frame: Up to 45 days post implantation
Population: The primary endpoint was wound occurrence within 45 days post implantation that required intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Xen Matrix AB: Subjects treated with Xen Matrix AB
  This group includes participants with a diagnosis of ventral or incisional midline hernia who have undergone the hernia surgical repair with the use of the XenMatrix AB.
Arm/Group | Xen Matrix AB
Number analyzed (Participants) | 75
Participants | 11

2. Secondary Outcome: Number of Participants With Wound Occurrences > 45 Days Post Implantation
Description: Wound occurrences was defined as surgical site infection, seroma, wound dehiscence, skin necrosis and fistulas requiring intervention.
Time Frame: Day 45 and up to 2 years post implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Xen Matrix AB
Number analyzed (Participants) | 75
Participants | 15

3. Secondary Outcome: Number of Participants With Hernia Recurrence Within 6 Months and 24 Months of Implantation Procedure
Time Frame: Within 6 months and 24 months of implantation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Xen Matrix AB
Number analyzed (Participants) | 75
Participants
  Within 6 Months | 0
  Within 24 Months | 4

4. Secondary Outcome: Number of Participants With Reoperation Due to Index Hernia Repair
Time Frame: 24 months post implantation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Xen Matrix AB
Number analyzed (Participants) | 75
Participants | 8

5. Secondary Outcome: Total Score on the Carolinas Comfort Scale (CCS) at Baseline, 1, 3, 6, 12, 18, and 24 Months Post Implantation Procedure
Description: The Carolinas Comfort Scale (CCS) quality of life questionnaire aimed for patients who have had hernia repair surgery. Symptoms in the CCS are rated by the participants on a scale of 0 to 5, with a score of 0 suggesting no symptoms and a score of 5, disabling symptoms. A lower score on the questionnaire compared to baseline would indicate a better outcome.
Time Frame: Baseline, 1, 3, 6, 12, 18, and 24 months post implantation procedure
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Subjects Treated With Xen Matrix AB
Number analyzed (Participants) | 75
Score on a scale
  Baseline: number analyzed (Participants) | 22
  Baseline | 1.6 (1.65)
  1 month: number analyzed (Participants) | 67
  1 month | 1.4 (1.42)
  3 months: number analyzed (Participants) | 65
  3 months | 1.2 (1.37)
  6 months: number analyzed (Participants) | 66
  6 months | 0.9 (1.18)
  12 months: number analyzed (Participants) | 59
  12 months | 0.8 (1.06)
  18 months: number analyzed (Participants) | 55
  18 months | 0.8 (1.15)
  24 months: number analyzed (Participants) | 58
  24 months | 0.6 (1.01)

6. Secondary Outcome: General Health Score on the Short Form 12 (SF-12) Questionnaire at Baseline, 1, 3, 6, 12, 18, and 24 Months Post Implantation.
Description: The Short Form 12 (SF-12) is a self-reported 12-item questionnaire that evaluates general health and well-being (overall quality of life of an individual). The SF-12 includes questions on physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100, with higher scores indicating better levels of functioning.
Time Frame: Baseline, 1, 3, 6, 12, 18, and 24 months post implantation
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Treated With Xen Matrix AB
Number analyzed (Participants) | 75
score on a scale
  Baseline: number analyzed (Participants) | 74
  Baseline | 47.7 (11.14)
  1 month: number analyzed (Participants) | 73
  1 month | 47.2 (10.30)
  3 months: number analyzed (Participants) | 67
  3 months | 48.6 (10.28)
  6 months: number analyzed (Participants) | 67
  6 months | 48.3 (9.77)
  12 months: number analyzed (Participants) | 59
  12 months | 48.3 (11.06)
  18 months: number analyzed (Participants) | 55
  18 months | 49.4 (9.17)
  24 months: number analyzed (Participants) | 58
  24 months | 47.9 (9.49)

7. Secondary Outcome: Number of Participants Who Returned to Work Post Implantation Procedure
Time Frame: Up to 2 years following implantation procedure
Population: The overall number of participants (21) for this endpoint reflects the number of participants who were employed at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Xen Matrix AB
Number analyzed (Participants) | 21
Participants | 17

8. Secondary Outcome: Duration of Participants Stay in Hospital Following Implantation Procedure
Time Frame: From index procedure day to discharge from hospital day
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Subjects Treated With Xen Matrix AB
Number analyzed (Participants) | 75
Days | 6.7 (6.13)

ADVERSE EVENTS:
Time Frame: From Day of index procedure up to 24 months post implantation procedure.
Arm/Group | Subjects Treated With Xen Matrix AB
All-Cause Mortality (participants affected / at risk) | 1/75
Serious Adverse Events (participants affected / at risk) | 31/75
Other Adverse Events (participants affected / at risk) | 55/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Treated With Xen Matrix AB (N=75)
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 3
Abdominal wall abscess (Infections and infestations) | 7
Bacteraemia (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Incision site infection (Infections and infestations) | 2
Necrotising fasciitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1
Iatrogenic injury (Injury, poisoning and procedural complications) | 3
Incisional hernia (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Pancreatic leak (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 9
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Treated With Xen Matrix AB (N=75)
Abdominal pain (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal wall abscess (Infections and infestations) | 7
Incision site cellulitis (Infections and infestations) | 5
Incision site infection (Infections and infestations) | 4
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 6
Anemia postoperative (Injury, poisoning and procedural complications) | 4
Iatronic injury (Injury, poisoning and procedural complications) | 4
Incisional hernia (Injury, poisoning and procedural complications) | 4
Postoperative ileus (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 9
Seroma (Injury, poisoning and procedural complications) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication of the principal results from any single-center experience within the study is not allowed until the preparation and publication of the multi-center results.

DOCUMENTS (2):
  • Study Protocol (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT02691962/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT02691962/SAP_001.pdf